CLINICAL TRIAL: NCT00490802
Title: Intranasal Oxytocin in the Treatment of Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evdokia Anagnostou (Individual)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor-Investigator, Evdokia Anagnostou, Clinician Scientist, Anagnostou, Evdokia, M.D.
Organization: Anagnostou, Evdokia, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-0230 0001 02 PS
Record Dates: First submitted 2007-06-22; First posted 2007-06-25 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Autism
Keywords: Autism; Treatment; Oxytocin; Adults; Autism Spectrum Disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Oxytocin (Experimental): Subjects were given 24 IU intranasal oxytocin twice daily, in the morning and afternoon for 6 weeks.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Subjects were given placebo twice daily, in the morning and afternoon for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Intranasal Oxytocin
  Other Names: Syntocinon
  Arms: Intranasal Oxytocin
Drug: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn whether or not the drug called oxytocin is helpful in improving mood and social functioning in adults with autism.

DETAILED DESCRIPTION:
Autism is a developmental disorder characterized by abnormalities in speech and communication, impaired social functioning, and repetitive behaviors and restricted interests. A number of researchers have suggested that the neuropeptide oxytocin may be implicated in the etiology of autism.

Given the likely possibility of dysregulated oxytocin in autism, the goal of this pilot study is to investigate the long-term therapeutic effects of oxytocin in the treatment of autism. One practical issue with oxytocin is that it does not exist in a pill form. Only the intravenous form is available in the United States and this form may or may not pass the blood-brain barrier. In addition, intravenous oxytocin is not practical for treatment studies. One alternative is intranasal oxytocin; this form of administration is known to pass the blood-brain barrier, and it is easy for participants to self-administer. Although not available in the United States, we are in the process of receiving an Investigational New Drug exemption for its use and can import it from Europe.

Thus, this pilot investigation will explore daily intranasal oxytocin in the treatment of autism. Also, there are very few, if any, outcome measures to assess social functioning in the "real world" in the context of clinical trials; yet, this is a major target for intervention, especially in autism. Thus, a final goal of this study will be to explore the use of Event Contingent Recording to index changes in social functioning and affect. Event Contingent Recording is a methodology developed by personality/social psychologists, which allows participants to report on symptoms, affect, and behavior close in time to experience. In addition, to enabling more sensitive assessments, this methodology allows for the assessment of more diverse (e.g., at home versus work) and more detailed measurements of mood and behavior.

Finally, a portion of this study aims to perform gene expression profiling using fresh whole blood to explore the molecular mechanisms underlying oxytocin therapy and oxytocin efficacy in adults with high functioning autism or Asperger's syndrome. The systemic effects of oxytocin therapy and the molecular basis for a positive treatment response to oxytocin are not well understood. An understanding of the former may help predict those persons who may suffer side-effects from treatment and the latter may help provide easily accessible peripheral biomarkers that could predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients 18 to 60 years of age.
2. Meet Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision. The diagnosis will be confirmed with Autism Diagnostic Interview-Revised and Autism Diagnostic Observation Schedule .
3. Have a Clinician's Global Impression-Severity score ≥ 4 (moderately ill) at Screening and Baseline.
4. If already receiving stable nonpharmacologic educational, behavioral, and/or dietary interventions, have continuous participation during the preceding 3 months prior to Screening and will not electively initiate new or modify ongoing interventions for the duration of the study.
5. Have normal physical examination and laboratory test results at Screening. If abnormal, the finding(s) must be deemed clinically insignificant by the Investigators.
6. The patient must be able to speak and understand English sufficiently to understand the nature of the study and to allow for the completion of all study assessments.
7. Have a normal Intelligence Quotient (>70) supported by the Wechsler Abbreviated Scales of Intelligence.

Exclusion Criteria:

1. Patients born prior to 35 weeks gestational age.
2. Patients with any primary psychiatric diagnosis other than autism at Screening: a history of attention deficit hyperactivity disorder, bipolar disorder, psychosis, posttraumatic stress disorder, schizophrenia, or major depressive disorder.
3. Patients with a medical history of neurological disease, including, but not limited to, epilepsy/seizure disorder (except simple febrile seizures), movement disorder, tuberous sclerosis, fragile X, and any other known genetic syndromes, or known abnormal magnetic resonance imaging/structural lesion of the brain.
4. Pregnant female patients.
5. Patients with a medical condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. Patients with evidence or history of malignancy or any significant hematological, endocrine, cardiovascular (including any rhythm disorder), respiratory, renal, hepatic, or gastrointestinal disease.
6. Patients taking psychoactive medication(s) (e.g., stimulants, antidepressants, antipsychotics, antiepileptics, anxiolytics, clonidine).
7. Patients who plan to initiate or change nonpharmacologic interventions during the course of the study.
8. Patients unable to tolerate venipuncture procedures for blood sampling.
9. Patients who, in the Investigator's opinion, might not be suitable for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2006-06; Primary Completion 2011-09 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Anagnostou E, Soorya L, Chaplin W, Bartz J, Halpern D, Wasserman S, Wang AT, Pepa L, Tanel N, Kushki A, Hollander E. Intranasal oxytocin versus placebo in the treatment of adults with autism spectrum disorders: a randomized controlled trial. Mol Autism. 2012 Dec 5;3(1):16. doi: 10.1186/2040-2392-3-16. PMID 23216716

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements in local media. Diagnosis was established using the Diagnostic and Statistical Manual, Fourth Edition criteria for an Autism Spectrum Disorder supported by the Autism Diagnostic Observation Schedule and the Autism Diagnostic Interview - Revised performed by research-reliable administrators.
Pre-assignment Details: This was a randomized, double-blind, placebo-controlled, parallel design trial of intranasal oxytocin versus placebo in adults with Autism Spectrum Disorder. As such, there were no participants excluded after enrollment but prior to assignment to groups.
Groups:
- Intranasal Oxytocin: Oxytocin : Intranasal Oxytocin
- Placebo: Placebo Comparator : Placebo Comparator
Period: Overall Study
Arm/Group | Intranasal Oxytocin | Placebo
Started | 10 | 9
Completed | 9 | 7
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Drug
  Placebo Comparator : Placebo Comparator
- Total: Total of all reporting groups
Arm/Group | Intranasal Oxytocin | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (12.7) | 32.9 (14.4) | 33.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impressions Scale - Improvement - Social
Description: The Clinical Global Impressions Scale - Improvement - Social is a well validated measure employing a 7-point scale of clinical global impression of improvement ( 1- very much improved, 2 - much improved, 3 - minimally improved, 4 - no change, 5 - minimally worse, 6 - much worse, 7 - very much worse) that the clinician fills out after considering all the available information on the participant including the parent history, the examination in clinic, reports from the school and other sources. Therefore the score is filtered through the judgment of the clinician evaluator.
  The Week 6 Improvement Ratings were used to categorize patients as clinically improved (≤2) or not (>2). Sixteen of the 19 patients (84%) had data at Week 6. For the remaining three subjects, Week 6 ratings were imputed using expectation-maximization methods and the earlier Clinical Global Impression ratings. In all three cases the imputed ratings were >2 and the patients were classified as not improved.
Time Frame: 6 Weeks
Measure: Number; unit: participants
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 10 | 9
participants | 3 | 1

2. Primary Outcome: Repetitive Behavior Scale - Revised
Description: The Repetitive Behavior Scale - Revised was developed to capture the breadth of repetitive behaviors that are specific to autism and is a parent report measure. In particular, it consists of 43-items that tap six repetitive behavior subtypes: Stereotyped, Self-injurious, Compulsive, Ritualistic, Sameness, and Restricted Interests.
  Two scores were calculated (higher-order vs. lower-order repetitive behaviors) in an effort to decrease the number of variables analyzed. This is based on previous factor analysis that produced these two factors: higher order (ritualistic, sameness, compulsive and restricted subscales) and lower order (stereotypy and self-injury).
  1. The higher order behaviors have 29 items that can be endorsed with a maximum score of 87 and a minimum score of 0
  2. The lower order behaviors have 14 items that can be endorsed, with a maximum score of 42 and a minimum score of 0
  In both cases, a lower score represents a positive response.
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 10 | 9
units on a scale
  Repetitive Behavior Scale - Revised - Higher Order | 17.7 (16.2) | 17.8 (13.3)
  Repetitive Behavior Scale - Revised -Lower Order | 2.4 (2.3) | 3.7 (2.6)

3. Primary Outcome: Diagnostic Analysis of Nonverbal Accuracy, Paralanguage Test
Description: The Diagnostic Analysis of Nonverbal Accuracy is a measure of emotion recognition across multiple modalities. It consists of five subtests: the Adult Facial Expression Test, the Child Facial Expression Test, the Adult Paralanguage Test, the Child Paralanguage Test, and the Adult Posture Test. The Diagnostic Analysis of Nonverbal Accuracy has established reliability and validity for children as young as 3 and adults as old as 100. The subtests of the test vary on four basic core emotions: happiness, sadness, anger, and fear, and the test provides measures of both high intensity and low intensity emotional reactions. We utilized both the Child Paralanguage and Adult Paralanguage Tests, therefore the minimum score that can be obtained is 0 and the maximum is 48. A higher score represents a positive response.
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 10 | 9
units on a scale | 30.5 (2.7) | 35.2 (4.7)

4. Secondary Outcome: Yale-Brown Obsessive-Compulsive Scale
Description: The Yale-Brown Obsessive-Compulsive Scale is a clinician-rated questionnaire measuring the time spent, distress, interference, resistance, and control in relation to obsessions and compulsions based on a 5-point scale. This scale has excellent reliability and validity and is used as the gold standard to measure treatment challenges in all Obsessive-Compulsive Disorder clinical trials. The Yale-Brown Obsessive-Compulsive Scale Compulsion Subscale has been shown to be a reliable and valid scale in Autism Spectrum Disorder, and in measuring change in treatment studies of autism. The minimum score that can be obtained is 0 and the maximum score is 20. A lower score represents a positive response.
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 10 | 9
units on a scale | 9.4 (2.9) | 8.1 (2.5)

5. Secondary Outcome: Social Responsiveness Scale
Description: The Social Responsiveness Scale has been developed to measure autism related symptoms and focuses more on social function than social cognition. The Social Responsiveness Scale has been modified for adults by and we have obtained permission to use the adult scale, although it is not commercially available yet. The Social Responsiveness Scale measures social behaviors such as social awareness, information processing, and social motivation and yields a quantitative score that has been useful in endophenotype studies of Autism Spectrum Disorder. The minimum score that can be obtained is a 0 and the maximum raw score for subscales is 66, maximum total raw score is 153. A lower score represents a positive response.
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 10 | 9
units on a scale | 111.4 (13.5) | 96.5 (13.0)

ADVERSE EVENTS:
Arm/Group | Intranasal Oxytocin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 9/10 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Oxytocin (N=10) | Placebo (N=9)
Irritability (Psychiatric disorders) | 1 | 0
Irritability (moderate) (Psychiatric disorders) | 1 | 0
Nasal congestion/allergy symptoms (Immune system disorders) | 2 | 0
Query absence seizures (Nervous system disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Leg shaking (Nervous system disorders) | 1 | 0
Increased energy (General disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Worsening tics (Nervous system disorders) | 0 | 1
Panic attack (moderate) (Psychiatric disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Small sample size resulted in baseline differences; short duration of study; didn't examine impact of other characteristics; short-half life in the blood; inactive ingredients not identical in placebo; no participant follow-up after study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No